CLINICAL TRIAL: NCT03224520
Title: Smoker-to-Smoker (S2S) Peer Marketing and Messaging to Disseminate Tobacco
Brief Title: Smoker-to-Smoker (S2S) Peer Marketing and Messaging to Disseminate Tobacco Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Massachusetts, Amherst (Other); Northwestern University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Rajani Sadasivam, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CDR-1603-34645; CDR160334645 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2017-06-21; First posted 2017-07-21 (Actual); Results first posted 2021-02-10 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Using a 2×2 factorial design, we will compare individually and collectively the enhancements (recruitment, use, and effectiveness) offered by the S2S functions over the standard version of Decide2Quit (online recruitment and standard CTHC), an active comparison group that was demonstrated to be effective in our previous trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fully enhanced (Experimental): Peer recruitment and recommender CTHC
  Interventions: Behavioral: Recommender CTHC; Other: Peer Recruitment
- Recommender CTHC only (Experimental): Recommender CTHC and standard online recruitment
  Interventions: Behavioral: Recommender CTHC; Other: Standard Online Recruitment
- Peer recruitment only (Experimental): Peer recruitment and standard CTHC
  Interventions: Behavioral: Standard CTHC; Other: Peer Recruitment
- Standard (Experimental): Standard online recruitment and standard CTHC
  Interventions: Behavioral: Standard CTHC; Other: Standard Online Recruitment

INTERVENTIONS:
Behavioral: Recommender CTHC — Enhanced Messaging
  Arms: Fully enhanced; Recommender CTHC only
Behavioral: Standard CTHC — Standard Messaging
  Arms: Peer recruitment only; Standard
Other: Peer Recruitment — Tools to facilitate smokers' recruiting their peers
  Arms: Fully enhanced; Peer recruitment only
Other: Standard Online Recruitment — Search Engine and Social Media Advertisements
  Arms: Recommender CTHC only; Standard

SUMMARY:
The research study, "Smoker-to-Smoker (S2S) Peer Marketing and Messaging to Disseminate Tobacco Interventions" will test two smoker-driven, social marketing innovations to recruit and engage smokers in Decide2Quit.org (Decide2Quit), which is an evidence-based, effective "Digital Intervention for Smoking Cessation".

DETAILED DESCRIPTION:
S2S has many innovations that are designed to utilize the power of peers and social networks for dissemination. These include: Peer recruitment: Tools to facilitate smokers' recruiting their peers to increase Decide2Quit access; and a recommender computer tailored health communication (recommender CTHC): a Complex machine learning algorithm (recommender systems) that uses smokers' feedback (explicit and implicit) in the current and prior studies to adapt its selection of messages to smokers.

Using a 2×2 factorial design, the study will compare individually and collectively the enhancements (recruitment, use, and effectiveness) offered by the S2S functions over the standard version of Decide2Quit (online recruitment and standard CTHC), an active comparison group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of Age or older
* Current smoker

Exclusion Criteria:

* Under 18 years of age
* Non-smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1487 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajani Sadasivam, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee DN, Faro JM, Stevens EM, Pbert L, Yang C, Sadasivam RS. Stopping use of E-cigarettes and smoking combustible cigarettes: findings from a large longitudinal digital smoking cessation intervention study in the United States. BMC Res Notes. 2024 Sep 27;17(1):276. doi: 10.1186/s13104-024-06939-w. PMID 39334264
- [Derived] Faro JM, Chen J, Flahive J, Nagawa CS, Orvek EA, Houston TK, Allison JJ, Person SD, Smith BM, Blok AC, Sadasivam RS. Effect of a Machine Learning Recommender System and Viral Peer Marketing Intervention on Smoking Cessation: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2250665. doi: 10.1001/jamanetworkopen.2022.50665. PMID 36633844
- [Derived] Chen J, Houston TK, Faro JM, Nagawa CS, Orvek EA, Blok AC, Allison JJ, Person SD, Smith BM, Sadasivam RS. Evaluating the use of a recommender system for selecting optimal messages for smoking cessation: patterns and effects of user-system engagement. BMC Public Health. 2021 Sep 26;21(1):1749. doi: 10.1186/s12889-021-11803-8. PMID 34563161
- [Derived] Faro JM, Nagawa CS, Orvek EA, Smith BM, Blok AC, Houston TK, Kamberi A, Allison JJ, Person SD, Sadasivam RS. Comparing recruitment strategies for a digital smoking cessation intervention: Technology-assisted peer recruitment, social media, ResearchMatch, and smokefree.gov. Contemp Clin Trials. 2021 Apr;103:106314. doi: 10.1016/j.cct.2021.106314. Epub 2021 Feb 8. PMID 33571687

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard
Started | 371 | 370 | 374 | 372
Completed | 205 | 207 | 190 | 199
Not Completed | 166 | 163 | 184 | 173

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard | Total
Number analyzed (Participants) | 371 | 370 | 374 | 372 | 1487
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 338 | 342 | 337 | 343 | 1360
  >=65 years | 33 | 28 | 37 | 29 | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 281 | 270 | 291 | 1101
  Male | 112 | 89 | 104 | 81 | 386
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 22 | 27 | 35 | 106
  Not Hispanic or Latino | 332 | 327 | 320 | 312 | 1291
  Unknown or Not Reported | 17 | 21 | 27 | 25 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 4 | 5 | 12
  Asian | 6 | 5 | 7 | 7 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2 | 0 | 4
  Black or African American | 43 | 42 | 37 | 38 | 160
  White | 295 | 293 | 288 | 291 | 1167
  More than one race | 11 | 12 | 16 | 15 | 54
  Unknown or Not Reported | 13 | 16 | 20 | 16 | 65
Number of Cigarettes Smoked per day [Count of Participants; unit: Participants]
  0 | 14 | 12 | 18 | 16 | 60
  >0 & <=10 Cigarettes | 121 | 112 | 117 | 108 | 458
  >10 & <=20 Cigarettes | 171 | 163 | 167 | 162 | 663
  >20 Cigarettes | 65 | 83 | 72 | 86 | 306
Smoking Status [Count of Participants; unit: Participants]
  Already quit | 48 | 56 | 61 | 67 | 232
  Thinking about quitting | 303 | 299 | 294 | 286 | 1182
  Not thinking about quitting | 17 | 10 | 17 | 18 | 62
  Missing | 3 | 5 | 2 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation
Description: Smoking cessation measured by the 7-day point prevalence question:
  Six month, 7-day point prevalence : Do you currently smoke cigarettes (smoked even 1 puff in the last 7 days)?
  * Yes
  * No
  * Don't know/not sure
  * Refused
Time Frame: At 6 months post registration
Measure: Count of Participants; unit: Participants
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard
Number analyzed (Participants) | 205 | 207 | 190 | 199
Participants
  Haven't smoked in last 7 days | 89 | 57 | 88 | 68
  Smoked in the last 7 days | 116 | 150 | 102 | 131

2. Secondary Outcome: Change in the Number of Cigarettes Smoked
Description: Calculated as: number of cigarettes smoked at six months minus the number of number of cigarettes smoked at baseline.
Time Frame: At 6 months post registration
Measure: Mean (Standard Deviation); unit: cigarettes a day
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard
Number analyzed (Participants) | 371 | 370 | 374 | 372
cigarettes a day | -9.60 (10.81) | -7.95 (10.15) | -10.63 (9.99) | -9.08 (11.41)

3. Secondary Outcome: Repeated Use of Decide2Quit Functions
Description: As measured by, an ordinal scale of number of Decide2Quit functions used after the first DISC visit (0: no functions used; 1: use of 1-2 functions, 2: > 2 functions used).
Time Frame: Throughout study (tracked for 6 months post registration)
Population: Analysis population limited to participants who visited Decide2Quit more than one time.
Measure: Count of Participants; unit: Participants
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard
Number analyzed (Participants) | 231 | 228 | 251 | 250
Participants
  No Use | 173 | 159 | 171 | 157
  1 or 2 Functions Used | 24 | 24 | 26 | 34
  Greater than 2 Functions Used | 34 | 45 | 54 | 59

4. Secondary Outcome: Recruitment of African Americans
Description: This is measured by the proportion of African Americans in each treatment arm
Time Frame: At Baseline Registration
Measure: Count of Participants; unit: Participants
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard
Number analyzed (Participants) | 371 | 370 | 374 | 372
Participants | 49 | 49 | 47 | 44

5. Secondary Outcome: Recruitment Time
Description: Calculated as: each individual participant's recruitment date minus the date of the first participant's registration. Based on this formula, the first participant will have a recruitment time of 0 days and the last participant could have a maximum recruitment time of 3 years (1095 days).
Time Frame: At Baseline Registration
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard
Number analyzed (Participants) | 371 | 369 | 373 | 371
days | 377.22 (135.80) | 379.29 (133.32) | 383.98 (136.84) | 367.28 (134.17)

ADVERSE EVENTS:
Description: Our study was an anonymous online smoking cessation intervention there were no risks to participants physical health associated with Decide2Quit. There was no possibility or risk for mortality associated with participation in our study. All-Cause Mortality, Serious, and Other (not including serious) Adverse Events were not monitored/assessed.
Arm/Group | Fully Enhanced | Recommender CTHC Only | Peer Recruitment Only | Standard
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03224520/Prot_SAP_000.pdf